CLINICAL TRIAL: NCT06152679
Title: Understanding the Patient Experience of Day-case Bladder Tumour Resection, and Prostate Resection or Enucleation: Qualitative Patient Interviews.
Brief Title: Day-case Endourology; Patient Experience
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: Royal Cornwall Hospitals Trust (Other); North Bristol NHS Trust (Other); Gloucestershire Hospitals NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other); Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 327246
Record Dates: First submitted 2023-11-21; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Bladder Cancer; Bladder Outflow Obstruction
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients who have undergone day-case bladder tumour resection or bladder outflow obstruction surgery (prostate resection or enucleation) within the past 6 weeks.
  Interventions: Other: None - qualitative interviews

INTERVENTIONS:
Other: None - qualitative interviews — Qualitative interviews with patients asking about their experience of day-case endourology.

SUMMARY:
A qualitative research study interviewing patients treated in hospitals across England. We will interview patients who have recently undergone one of the following operations as a day-case; transurethral bladder tumour resection (TURBT), transurethral resection of prostate (TURP) or transurethral enucleation of the prostate (TUEP). We are interested to find out about the experience for patients who go home on the day of surgery after they have had one of these operations. We hope that the findings will tell us about how to improve the experience for patients in future.

Patients undergoing day-case surgery at a range of different hospitals from across England with varying day-case rates will be interviewed. Hospitals in large city and more rural areas will be included. Interviews are anticipated to take place over a six month period. The study will end when "saturation" is achieved, whereby no new themes are identified through interviews. Saturation will be sought for each individual operation of interest.

DETAILED DESCRIPTION:
Safe day-case surgery pathways offer to reduce pressure on hospitals by avoiding overnight inpatient admission. This is particularly relevant given the intense pressures on hospital resources in the United Kingdom. Urological surgery includes a number of frequently performed operations for which safe day-case surgery pathways have been demonstrated, but for which day surgery is routine widespread routine practice. These include bladder tumour resection (TURBT), and prostate resection or enucleation using diathermy or laser (TURP and TUEP). All of these operation types involve endoscopic access to the bladder via the urethra, and do not involve skin incisions. They can be performed under general or spinal anaesthesia.

For 12 months from December 2021, the national average day-case rate for transurethral resection of bladder tumour In England was 21.1%, and ranged from 0% to 87.3% at different hospitals, with an interquartile range (IQR) of 10.5% to 37.7%, and 23,071 cases performed in total. For bladder outflow obstruction surgery the median day-case rate was 7.7% (range 0% to 82.4%, IQR 4.4% to 19.1%, 18,912 cases), and this includes TURP and TUEP. This demonstrates that for these common operations there is significant variation in practice across England.

The Getting It Right First Time (GIRFT) Urology programme advocates for a "day-case by default" approach to TURBT, and that day-case surgery should ideally be offered for prostate resection and enucleation. As well as reducing pressure on inpatient services, greater day-case adoption offers to reduce financial costs, shorten waiting lists by allowing greater access to day-case theatres away from the acute hospital, and reduce environmental impact by adopting a less resource-intensive approach. It also offers a more standardised patient experience, however we do not understand a great deal about the lived patient experience after discharge.

National day-case rates for of TURBT, and bladder outflow obstruction surgery using TURP or TUEP, have increased over the past five years. Many hospitals have well-established pathways, whilst others are newly adopting this approach, or not yet adopting day-case surgery for these operation types at all. There is an opportunity to understand the patient experience of different day-case surgery pathways for these operations of interest, so that we might understand factors contributing to a favourable or unfavourable experience. This knowledge could inform future day-case pathway development and modification is a way that is more acceptable for patients.

To explore this area, we intend to perform qualitative research involving patients. We will interview patients who were treated at a range of different hospitals with differing day-case performances.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or more
* Experienced day-case TURBT, TURP or TUEP within the past 6 weeks
* Willing and able to provide informed consent
* English speaking

Exclusion Criteria:

* Experienced surgery that was not performed as a day-case

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have recently undergone day-case transurethral resection of bladder tumour (TURBT), transurethral resection of prostate (TURP), or transurethral enucleation of the prostate (TUEP) at an NHS hospital in England.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Patient description of their experience | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Devon University Healthcare NHS Foundation Trust, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
None. Only anonymised quotes will be used in published study write-up.

DOCUMENTS (1):
  • Study Protocol (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT06152679/Prot_000.pdf